CLINICAL TRIAL: NCT04675086
Title: A Randomized, Open-Label Study of the Efficacy and Safety of Aralast NP, an Alpha-1 Antitrypsin Infusion Therapy With Antiviral Treatment and Standard of Care Versus Antiviral Treatment With Standard of Care in Hospitalized Patients With Pneumonia and COVID-19 Infection
Brief Title: Aralast NP With Antiviral Treatment and Standard of Care Versus Antiviral Treatment With Standard of Care in Hospitalized Patients With Pneumonia and COVID-19 Infection
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative Decision
Sponsor: Blessing Corporate Services, Inc (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR-2020-103188
Record Dates: First submitted 2020-11-25; First posted 2020-12-19 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Pneumonia, Viral
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — alpha 1-Antitrypsin; Antiviral Agents; remdesivir

STUDY DESIGN:
Intervention Model Description: Randomized with 1:1 ratio to the high dose of Aralast NP infusion therapy plus antiviral and standard of care versus antiviral therapy and standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aralast NP + Antiviral Treatment + Standard of Care (Experimental): The investigational product is alpha1-proteinase inhibitor, administered as a loading dose of 120mg/kg/body weight intravenous infusion on the first day, and then 60mg/kg/BW intravenous infusion on Days 3, 5, 7 and 9. Booster infusion of 120 mg/kg/BWon Day 17.
  The Antiviral treatment is Remdesivir. For patients not requiring invasive mechanical ventilation and/or ECMO, the recommended total treatment duration is 5 days. If a patient does not demonstrate clinical improvement, treatment may be extended for up to 5 additional days for a total treatment duration of up to 10 days. Recommended dosage in adults and pediatric patients 12 years of age and older and weighing at least 40 kg: a single loading dose of Remdesivir 200 mg on Day 1 followed by once-daily maintenance doses of Remdesivir 100 mg from Day 2 infused over 30 to 120 minutes
  Standard of Care treatments are at the investigator's discretion based on best practices.
  Interventions: Drug: alpha1-proteinase inhibitor; Drug: Antiviral Agents
- Antiviral Treatment + Standard of Care (Active Comparator): The Antiviral treatment is Remdesivir. For patients not requiring invasive mechanical ventilation and/or ECMO, the recommended total treatment duration is 5 days. If a patient does not demonstrate clinical improvement, treatment may be extended for up to 5 additional days for a total treatment duration of up to 10 days. Recommended dosage in adults and pediatric patients 12 years of age and older and weighing at least 40 kg: a single loading dose of Remdesivir 200 mg on Day 1 followed by once-daily maintenance doses of Remdesivir 100 mg from Day 2 infused over 30 to 120 minutes
  Standard of Care treatments are at the investigator's discretion based on best practices.
  Interventions: Drug: Antiviral Agents

INTERVENTIONS:
Drug: alpha1-proteinase inhibitor — Alpha1-Proteinase Inhibitor (Human), AralastÔ, is a sterile, stable, lyophilized preparation of purified human alpha1-proteinase inhibitor (a1-PI), also known as alpha1-antitrypsin.
  Other Names: Aralast NP
  Arms: Aralast NP + Antiviral Treatment + Standard of Care
Drug: Antiviral Agents — a SARS-CoV-2 nucleotide analog RNA polymerase inhibitor indicated for adults and pediatric patients (12 years of age and older and weighing at least 40 kg) for the treatment of coronavirus disease 2019 (COVID-19) requiring hospitalization
  Other Names: Remdesivir

SUMMARY:
This is a Randomized, Open-Label Study of the Efficacy and Safety of Aralast NP Infusion Therapy with Antiviral Treatment and standard of care versus Antiviral Treatment and standard of care (control group) in Hospitalized Patients with Pneumonia and COVID-19 Infection.

DETAILED DESCRIPTION:
Approximately 20 subjects in total will be randomized with 1:1 ratio to the high dose of Aralast NP infusion therapy plus antiviral and standard of care versus antiviral therapy and standard of care.

Each subject will participate in the study for 24 days and have one safety follow-up phone call at 30 days. Active treatment will last 17 days, subject will be dosed on Days 1, 3, 5, 7, 9 and have a final booster infusion on Day 17. If the subject is discharged from hospital, any remaining infusions and assessments will be conducted via outpatient clinic visit or home health visit. Subjects will have an in-person visit (hospital or clinic) on Day 24 for a CT scan and follow-up assessment.

Efficacy will be evaluated by measuring the duration of new non-invasive ventilation or high flow oxygen used. Additional endpoints include clinical status, cytokine levels, oxygen requirements, SOFA scores, risk of coagulopathy, need for Vasopressors, mortality during the treatment period, PK samples, average days spent in the hospital/ICU, and number of days without a fever.

ELIGIBILITY:
Inclusion Criteria

1. Subject will sign and date an informed consent form.
2. Hospitalized subjects will be 18 years of age or older.
3. Lab confirmed positive for COVID-19 within 72 hours prior to randomization.
4. Subjects with COVID-19 with evidence of pneumonia (diagnosed by a chest x-ray) on supplemental oxygen or non-invasive ventilation with PO2/FiO2 ratio less than 300.
5. Subject must have one of the following elevated inflammatory markers: C-reactive protein >40mg/L; D-Dimers > 250ng/mL DDU or >0.5mcg/mL FEU; Ferritin >400ng/mL; LDH >300U/L.

Exclusion Criteria

1. Subject is on mechanical ventilation at time of screening.
2. Subject is not expected to survive greater than 48 hours from screening based on PI judgement.
3. Prior or current treatment with anti-IL-6, anti-IL-6 R antagonist or JAK inhibitors.
4. Subject is on immunosuppressive agents, with the exception of corticosteroids for severe COVID-19 patients at the discretion of the PI.
5. Subject is currently participating in a trial for any other investigational drug.
6. Subject is on another plasma derived product or has received plasma or blood products within the last 48 hours.
7. Subject is pregnant or breastfeeding.
8. The subject, or the next of kin/power of attorney are not able to give the proper informed consent.
9. The subject has a known IgA deficiency with anti-IgA antibodies.
10. Subject has a known Alpha-1 Antitrypsin Deficiency.
11. Subject has antibodies against alpha-1 proteinase inhibitor
12. Subject has renal, liver or multisystem organ failure
13. Subject has known history of hypersensitivity following infusions of human blood or blood components (eg, human immunoglobulins or human albumin).
14. Positive serological test for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Duration of new non-invasive ventilation or high flow oxygen use (measured by days) | 365 Days

SECONDARY OUTCOMES:
Clinical status on a 7-point ordinal scale (from 1=death to 7=not hospitalized | 1 Year
The percentage change in cytokine levels from screening through day 10, Day 17 and Day 24 | 10 Days, 17 Days, & 24 Days
The percentage change in oxygen requirements including PEEP and FiO2 from screening through day 10. | 10 Days
The percentage of subjects that required mechanical ventilation during the treatment period. | 1 Year
The percent of patients with a SOFA score between 0-6 during treatment period. | 1 Year
The percent of mortality during the treatment period. | 1 Year
Evaluate the need, dosage and duration of vasopressors (number of days and average daily dose). | 1 Year
Number of Days fever free (defined by temperature of <100°F (oral) for 24 hours) | 1 Year
To evaluate the average number of days in the ICU | 1 Year
To evaluate the average number of days in the hospital | 1 Year
To evaluate the number of days with a PO2/FiO2 <300 or other parameters decided on with oxygen | 1 Year
The risk of coagulopathy by measuring Prothrombin time & Partial Thromboplastin time | 1 Year
The risk of coagulopathy by measuring D-Dimer | 1 Year
The risk of coagulopathy by measuring Platelet Counts | 1 Year

OTHER OUTCOMES:
The percentage of patients with lung fibrosis or worsening of lung fibrosis from screening to Day 10 and Day 24 (as assessed by CT). | 10 Days, 17 Days, & 24 Days
Maximal inspiratory pressure (MIP) at Day 10, Day 17 and Day 24. | 10 Days, 17 Days, & 24 Days
Maximal expiratory pressure (MEP) at Day 10, Day 17, and Day 24. | 10 Days, 17 Days, & 24 Days
Muscle strength assessment at Day 10, Day 17 and Day 24. | 10 Days, 17 Days, & 24 Days
Correlation between plasma exposure of Aralast NP (Pharmacokinetics) and the other listed clinical endpoints at Days 1, 3, 5, 7, 9 and 17. | 1 Day, 3 Days, 5 Days, 7 Days, 9 Days, & 17 Days
  Pharmacokinetics of Aralast NP levels will be drawn to determine if there is a correlation between that and the other endpoints listed above.
Correlation between plasma exposure of Aralast NP (Pharmacokinetics) and biomarker endpoints (Pharmacodynamics) at Days 1, 6, 10 and 17 | 1 Day, 6 Days, 10 Days, & 17 Days

CONTACTS AND LOCATIONS:
Overall Officials: Humam Farah, MD, Principal Investigator — Employee
Locations (1):
- Blessing Corporate Services, Inc, Hannibal, Missouri, United States

IPD SHARING:
Plan to Share IPD: No